CLINICAL TRIAL: NCT02943278
Title: Sleep Therapy for Insomnia and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Leslie Swanson, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00112746
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Depression; Insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Hygiene Group (Placebo Comparator): Participants assigned to the sleep hygiene group you have 1 session with a clinician to learn about different things they can do to improve their sleep.
  Interventions: Behavioral: Sleep Hygiene
- Intensive Sleep Retraining Group (Active Comparator): Participants assigned to this group will spend just over 1 day at our sleep lab, starting around your usual bedtime and ending the following day. Over a 20 hour period participants will complete a sleep retraining session, which involves an opportunity to fall asleep every 30 minutes; we will wake the participant up after a few minutes if they fall asleep.
  Interventions: Behavioral: Intensive Sleep Retraining

INTERVENTIONS:
Behavioral: Intensive Sleep Retraining — Participants in this group you will spend just over 1 day at our sleep lab, starting around their usual bedtime and ending the following day. Over a 20 hour period participants will complete a sleep retraining session, which involves an opportunity to fall asleep every 30 minutes; we will wake participants up after a few minutes if they fall asleep.
  Arms: Intensive Sleep Retraining Group
Behavioral: Sleep Hygiene — Participants in this group will complete one session with a clinician focused on psychoeducation regarding sleep positive practices.
  Arms: Sleep Hygiene Group

SUMMARY:
In this study we are testing 2 different forms of sleep therapy to help people with insomnia and depression. As part of the study, you receive 1 of these 2 sleep therapies. We want to see how these sleep therapies help insomnia in people with depression.

DETAILED DESCRIPTION:
The first group is the sleep hygiene group. If you are assigned to the sleep hygiene group you have 1 session with a clinician to learn about different things you can do to improve your sleep.

The second group is the intensive sleep retraining group. If you are in this group you will spend about 1 day at our sleep lab, starting around your usual bedtime and ending the following day. Over a 20 hour period you will complete a sleep retraining session, which involves an opportunity to fall asleep every 30 minutes; we will wake you after a few minutes if you fall asleep.

For both groups, after the treatment session, you will complete questionnaires online and talk with a study clinician who will ask you questions about your mood every two weeks for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing depression
* Experiencing chronic insomnia
* Have been taking an antidepressant medication at a stable dose for at least 8 weeks, and willing to stay on a stable dose for the duration of the study. This medication must be prescribed by a doctor at the University of Michigan. OR not taking any antidepressants and you do not plan to start taking any antidepressants over the next 9 weeks.

Exclusion Criteria:

* Have psychiatric conditions or sleep disorders other than depression or insomnia
* Have a chronic medical condition that could negatively affect your sleep or mood
* Are currently receiving treatment for insomnia (such as prescription or over-the-counter medications, or other therapies)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Score of the Hamilton Depression Rating Scale at 8 weeks | 8 weeks after administration of intervention
  Clinician-rated depression symptom severity measure

SECONDARY OUTCOMES:
Change from Baseline Score of the Insomnia Severity Index at 8 weeks | 8 weeks after administration of intervention
  Self report measure of insomnia symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Swanson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No